CLINICAL TRIAL: NCT01059877
Title: Assessing the Effect of 1072nm Infrared (IR) Phototherapy on the Behavioral and Cognitive Symptoms Associated With Early and Mid-stage Dementia: a Randomized Placebo-controlled Clinical Trial.
Brief Title: Efficacy of 1072nm Infrared Stimulation on Executive Functioning in Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quietmind Foundation (Other)
Collaborators: Maculume Ltd. (Industry)
Responsible Party: Principal Investigator, Marvin H. Berman, Ph.D., clinical trial coordinator, Quietmind Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QMF-MID12610
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Dementia
Keywords: dementia alzheimers frontotemporal lyme,; lewy body cognitive impairment
MeSH Terms: conditions — Dementia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Small placebo controlled randomized trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1072nm Infrared Photobiomodulation (Active Comparator): Received treatment for dementia with transcranial 1072nm infrared light stimulation.
  Interventions: Device: 1072nm infrared Photobiomodulation
- Placebo (Placebo Comparator): Placebo device simulated transcranial photobiomodulation
  Interventions: Device: Photobiomodulation SIMULATED

INTERVENTIONS:
Device: 1072nm infrared Photobiomodulation — 1072nm infrared light delivering 2.6 Joules (2.6J)/sq cm over a 6 minute treatment period.
  Other Names: Photobiomodulation, Low-level LED Light Stimulation
  Arms: 1072nm Infrared Photobiomodulation
Device: Photobiomodulation SIMULATED — Device mounted and procedure followed but with no stimulation.
  Arms: Placebo

SUMMARY:
This study will employ a double-blind, placebo-controlled approach to assess the effect of 1072nm infrared (IR) phototherapy on the behavioral and cognitive symptoms associated with early and mid-stage dementia.

DETAILED DESCRIPTION:
What hypotheses are you testing?

We are seeking to determine if the provision of brief, repeated exposure to 1072nm infrared stimulation of the cortex surface improves cognitive and behavioral functioning as indicated by normalization of EEG activity, increased cerebral oxygenation and demonstrated improvement on standardized neuropsychological measures.

Intensive near infrared stimulation has been shown to be effective in accelerating healing of injuries and functional modification including increasing blood flow and perfusion. Dementia research has suggested that hypoperfusion is a significant underlying mechanism in the progression of dementia. Infrared spectroscopy has been shown effective in the non-invasive measurement of changes in cerebral oxygenation and perfusion. This study therefore seeks to explore whether the increasing of regional cerebral perfusion and oxygenation using infrared light stimulation will result in improved cognitive and behavioral functioning.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50 - 85 years.
* Have established cognitive impairment, Mini Mental Status Examination (MMSE) score between 15- 25 (from a possible score of 30).
* Generally healthy otherwise as indicated by recent physical examination.
* Have a caregiver/informant who has cared for the patient at least 5 days a week and is willing to attend study visits and provide information about the patient.
* If taking any psychotropic medication should have been stable for the previous 3 months.
* Must have had B12, folic acid, full blood count and ferritin screen within the previous 6 months or be on B12 and/or folic acid replacement.

Exclusion Criteria:

* Uncontrolled or unstable chronic illness, e.g., hypertension, chronic obstructive pulmonary disease (COPD).
* Diagnosed actively growing intracranial pathology (tumors etc).
* An associated psychotic illness.
* Misusing illegal substances or alcohol.
* On regular systemic steroids or anti-metabolites.
* Systemic malignancies and/or space occupying lesions in the brain.
* Not fluent in English.
* Depressed as assessed by Beck Depression Inventory score.
* Epilepsy.
* Lacking the capacity to give informed consent.
* Previous history of stroke or heart attack.
* History of aggression or violence.
* Inability to travel to the research venue for multiple assessments.
* A history of major psychiatric illness, seizure disorder, or physical illness that would compromise their participation in a daily treatment regimen.
* A participant may be disqualified if their performance is above the normative mean or below the lowest interpretable score of neuropsychological tests provided during the initial assessment (see #6, Sources of research material obtained from study participants, below).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marvin H Berman, Ph.D, Principal Investigator — Quietmind Foundation
Locations (1):
- Quietmind Foundation, Plymouth Meeting, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berman MH, Halper JP, Nichols TW, Jarrett H, Lundy A, Huang JH. Photobiomodulation with Near Infrared Light Helmet in a Pilot, Placebo Controlled Clinical Trial in Dementia Patients Testing Memory and Cognition. J Neurol Neurosci. 2017;8(1):176. doi: 10.21767/2171-6625.1000176. Epub 2017 Feb 28. PMID 28593105

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: received actual tx
- Placebo Group: received placebo tx
Period: Overall Study
Arm/Group | Treatment Group | Placebo Group
Started | 6 | 5
Completed | 6 | 3
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Mean (Full Range); unit: years] | 80 [74 to 89] | 84 [76 to 96] | 81 [74 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 1 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 3 | 9
Delayed word recall [Mean (Full Range); unit: units on a scale] — Delayed Word Recall is a subscale of the Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog), a measure of cognitive impairment. Higher scores indicate greater impairment. Range: 0-10.
  units on a scale | 0.50 [0 to 1] | 1.33 [0 to 4] | 0.798 [0 to 4]
Trail making A [Mean (Full Range); unit: errors at task] — The Trail Making Test (TMT) is used to investigate deficits in cognitive processing speed and executive function. Part A consists of 25 circles on a piece of paper with the numbers 1-25 in random order in the circles. The patient starts with number one and draws a line from that circle to the circle with number two, etc. to number 25. More errors indicate poorer performance.
  errors at task | 0.83 [0 to 5] | 9.00 [3 to 14] | 3.56 [0 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer Disease Assessment Scale-Cognitive (ADAS-Cog) Delayed Word Recall.
Description: Delayed Word Recall is a subscale of the Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog), a measure of cognitive impairment. Higher scores indicate greater impairment. Range: 0-10. Measures were taken within 72 hours of the first day of treatment and within 72 hours following the 28th day of treatment. Outcome measure was calculated by subtracting pretest from post test ADAS-Cog measurements.
Time Frame: Post-tx (total intervention period = 28 days) scores to be compared to baseline scores.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment Group | Placebo Group
Number analyzed (Participants) | 6 | 3
units on a scale | 3.17 [2 to 4] | 3 [3 to 3]

ADVERSE EVENTS:
Time Frame: Course of study, approx. 6 months
Arm/Group | Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No